CLINICAL TRIAL: NCT02655757
Title: Effect of Sitagliptin on Progression of Coronary Intermediate Lesion in Patients With Coronary Heart Disease Complicated With Type 2 Diabetes
Brief Title: Effect of Sitagliptin on Progression of Coronary Intermediate Lesion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Li Bo (Other)
Responsible Party: Sponsor-Investigator, Li Bo, Director, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 301_xnk
Record Dates: First submitted 2015-12-27; First posted 2016-01-14 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Atherosclerosis; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Atherosclerosis; Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sitagliptin (Active Comparator): Sitagliptin 100mg QD
  Interventions: Drug: Sitagliptin
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sitagliptin — 5 mg, 1 tablet per day for 12 months
  Other Names: JANUVIA
  Arms: Sitagliptin
Drug: Placebo — Placebo,1 tablet per day for 12 months
  Arms: Placebo

SUMMARY:
This study was to investigate the Effect of Sitagliptin, a dipeptidyl peptidase-4 inhibitor, on Progression of Coronary Intermediate Lesion.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18, < 80 years old, with type 2 diabetes mellitus and angiographically proven Coronary Intermediate Lesion.

Exclusion Criteria:

* Allergy or hypersensitivity to any of the drug's components.
* Severe liver failure, moderate or severe kidney failure
* Malignant disease.
* Active infectious disease.
* Pregnancy or breastfeeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-12; Primary Completion 2017-02-02 (Actual); Study Completion 2017-03-10 (Actual)

PRIMARY OUTCOMES:
Changes in late lumen loss of target lesion | Changes from baseline in late lumen loss of target lesion at 12 months
  A coronary intermediate lesion in Patients with coronary heart disease complicated with Type 2 Diabetes was measure with 3D QCA(3D Quantitative Coronary Angiography). To measure the changes in target lumen at 12 months.

SECONDARY OUTCOMES:
Incidence rate of MACE | Incidence rate of MACE from baseline to 12 months
  MACE include composite of death, myocardial infarction, or target-vessel revascularization.

CONTACTS AND LOCATIONS:
Overall Officials: Chen yundai, MD, Principal Investigator — The General Hospital of PLA
Locations (1):
- The General Hospital of PLA, Beijing, Beijing Municipality, China